CLINICAL TRIAL: NCT04366817
Title: Psychological Impact of the Lockdown on Patients Giving Birth During the COVID-19 Epidemic
Brief Title: Psychological Impact of the Lockdown on Patients Giving Birth During the COVID-19 Epidemic Short Title : Isolement and Childbirth: Psychological Impact
Acronym: COVMUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: APHP200471
Record Dates: First submitted 2020-04-20; First posted 2020-04-29 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Post Partum Depression
Keywords: COVID-19 - Sars-CoV2; quarantine Depression; Postpartum
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- women in postpartum period (Experimental)
  Interventions: Behavioral: psychological assessment

INTERVENTIONS:
Behavioral: psychological assessment — psychological assessment at D10-12 and 6-8 weeks : Scheduled telephone interview using the assessment scales (EPDS, PPQ, MIBS, DAS-16) on D10-D12 and 6-8 weeks postpartum with a psychologist

SUMMARY:
The COVID-19 epidemic has a major impact on the organization of hospital structures as a whole. Regarding the functioning of the Maternities, it was decided by the three Maternities of AP-HP. Sorbonne University of the Pitié-Salpêtrière, Trousseau and Tenon sites, from March 20, 2020 to no longer authorize visits during the stay of mothers following childbirth. This prohibition has also been extended to spouses. This measure was guided by a concern to protect both the patients, their newborn and the entire staff of the aftermath.

The period surrounding a birth is a period of strong emotional impact with an incidence of postpartum depression estimated at 15% in the general population (1). The separation of women from their spouses during this period could expose them to greater psychological vulnerability. In addition, when they return home, the patients will be isolated from their relatives due to the quarantine, which is an additional risk factor for postpartum depression. The teams of the three maternity units of AP-HP. Sorbonne University have organized themselves to be able to respond to situations of mental vulnerability during their stay with the intervention of maternity psychologists and psychiatrists and child psychiatrists as is done in the treatment usual charge. In addition, anticipating situations of greater vulnerability linked to the health crisis, the Maternity teams decided to set up a follow-up of patients after their return home through a telephone interview with psychologists or student psychologists in Master at D10 - D12 and 6-8 weeks postpartum in order to identify patients at increased risk of postpartum depression and to set up appropriate management if necessary for these patients.

We therefore propose through this project to describe the consequences of this separation from the spouse during the postpartum stay and then with the family after returning home within the context of quarantine by assessing the incidence of post-partum depression during this sanitary crisis. A telephone interview of all the patients will be proposed on D10 - D12 and at 6-8 weeks postpartum using specific questionnaire to calculate a score of depression. This early identification will allow the establishment of an adapted psychological follow-up.

DETAILED DESCRIPTION:
The main objective of this study is to assess the emotional impact of the separation of women from their spouses following childbirth and their family isolation when returning home within the context of quarantine due to the COVID epidemic.

The secondary objectives are:

1. To identify the factors of greatest vulnerability or resilience of the patients in the immediate postpartum period (6-8 weeks after delivery).
2. To evaluate the impact of quarantine on the couples (DAS-16 scale), the experience of childbirth (PPQ scale), mother-child interactions (MIBS) at D10-D12 postpartum and at 6-8 weeks postpartum.
3. Recording of all interviews allowing a qualitative study of the verbatim by the use of N-Vivo software allowing the analysis of unstructured and qualitative data.

The primary endpoint will be the proportion of patients with postpartum depression defined by EPDS score >12 at D10-12 and 6-8 weeks postpartum. The EPDS relies on 10 specific items which allows the calculation of a depression score. A threshold > 12 is used in research to define the existence of depressive symptoms. For research, the score can be used as a continuous variable or in class with the threshold value 12.

The secondary end points will be:

1. to study factors of greatest vulnerability or resilience of the patients will be studied:

   * Socio-economic data
   * maternal or fetal pathology during previous pregnancies
   * associated pregnancy pathology
   * Maternal psychologic history
2. to describe the impact on the couple (DAS-16 scale), the experience of childbirth (PPQ scale), mother-child interactions (MIBS):

   * Dyadic Adjustment scale 16 (DAS-16). Revised scale was developed to assess dyadic adjustment in marriage.
   * Perinatal Posttraumatic Stress Disorder Questionnaire (PPQ). This self-questionnaire makes it possible to assess the post-traumatic reactions of parents faced with the birth of a child presenting a high perinatal risk.
   * Mother-to-Infant Bonding Scale (MIBS): Auto questionnaire, initially developed with a view to researching disturbances in maternal feelings towards the newborn. The scores range from 0 to 24, a high score being in favor of a mother-child bond disorder.
3. Automated psycho-linguistic analysis of the interviews using the N Vivo software. This software allows an automated study of the verbatim allowing a qualitative analysis of prosody and to identify emotional profiles and thus to identify situations of anxiety, stress and depression.

The study population will consist of patients with delivery of a child and:

* Singleton pregnancy
* Alive child without hospitalization of the child in NICU
* Patient speaking and understanding French
* Major patient

Duration of inclusion will be 2 months The Inclusion visit will take place during hospitalization in post-partum units, signed consent informed will be collected by a qualified person (medical doctor or midwife) before inclusion. Each week, these forms will be sent to the study psychologist referent in each of the 3 Maternity units.

Research follow-up visits:

Scheduled telephone interview using the assessment scales described above on D10-D12 and 6-8 weeks postpartum with a psychologist or an M2 psychology student under the responsibility of a maternity psychologist. A reminder system is provided by sending an SMS / email 48 hours before the scheduled call. In the event of a missed call, a re-call is scheduled on the same day or the next day (the SMS / email sent to patients indicates this reminder mode in the event of unavailability during the first call).

During this call, a semi-structured interview is carried out with EPDS score, DAS-16 scale, PPQ and MIBS questionnaire, and a recording for analysis of unstructured and qualitative data.

When EPDS score> 12: proposal for psychological follow-up in accordance with current standard of care in the event of postpartum depression.

For scores <12, the possibility of a further interview with a psychologist, apart from the study, is formulated.

Telephone interview at 6-8 weeks with psychologist including, as previously described, a semi-structured interview with EPDS score, DAS-16 scale and MIBS questionnaire and a recording for analysis of unstructured and qualitative data When EPDS score> 12: proposal for psychological follow-up in accordance with current standard of care in the event of postpartum depression.

For scores <12, the possibility of a further interview with a psychologist is formulated.

The patients were informed of the recording of the calls. In case of refusal, the calls are not recorded and only the semi-structured interview is carried out with EPDS score and DAS-16 scale and PPQ and MIBS questionnaire.

Sample size justification The inclusion of 452 women will allow to detect at least a 5 points change in the proportion of postpartum depression during COVID pandemic period compared to the expected/usual proportion of 15% (15 vs. 20%) with 80% of power, considering two-sided alpha risk of 5% and 5% of dropout.

ELIGIBILITY:
Inclusion Criteria:

-- Single pregnancy

* Birth of a child living without hospitalisation of the child in Neonatology (outside the accommodation of the newborn in Neonatology for maternal reasons)
* Patient speaks and understands French
* Patient affiliated to social security
* Major patient
* Written consent or nonopposition if retrospectif inclusion

Exclusion Criteria:

- Protected patient or patient unable to give consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2021-02-17 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with postpartum depression defined by an EPDS score >12 | Between week 6 and week 8
  assess the emotional impact of women's separation from their partners following childbirth and then their family isolation when they return home in the context of the health crisis linked to the COVID-19 epidemic
Proportion of patients with postpartum depression defined by an EPDS score >12 | Between day 10 and day 12
  assess the emotional impact of women's separation from their partners following childbirth and then their family isolation when they return home in the context of the health crisis linked to the COVID-19 epidemic

SECONDARY OUTCOMES:
Socio-demographic data | Between day 1 and day 5
Occurrence of a maternal or fetal pathology in a previous pregnancy | Between day 1 and day 5
Pregnant maternal pathology (hypertension, diabetes, threat of premature delivery) | Between day 1 and day 5
Presence of psycological maternal risk factor | Between day 1 and day 5
  as above, maternal psychological history as vulnerability factor included : history of perinatal loss, IMG, history of post partum depression.
Dyadic adjustment scale 16 (DAS-16) | Between day 10 and day 12 and at between week 6 and week 8
Perinatal post traumatic stress disorder questionnaire (PPQ scale) | Between day 10 and day 12
Mother to infant bonding scale (MIBS) autoquestionnaire | Between day 10 and day 12 and at between week 6 and week 8
Measure Qualitative Interviews by Grounded theory | Week 14
  Participants will be asked open-ended questions about their post-partum experience in the context of COVID-19 epidemic lockdown. The interviews will be transcribed and tagged with codes which have been extracted from the data. As more data is collected codes can be regrouped into concepts and then categories. These categories are the basis of the "theory model" that emerge from the narrative of the patients.
  The verbatim of the interview will be analyzed using NVIVO software which allows a grounded theory approach.
  Using software package as Nvivo (Hutchison, 2010) with automatic analysis of the verbatim to extract codes and concepts provides a transparent account of the data and enhance study validity.
  Verbatim are download in the software, that extract repeated lexical fields the categories from the mother's narrative.
  As this is a qualitative study, there are no expected outcomes. Outcomes will be determined by the themes that arise from the post-partum interview process.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Marie JOUANNIC, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service médecine foetale-Hôpital Trousseau, Paris, France

REFERENCES:
- [Derived] Viaux-Savelon S, Maurice P, Rousseau A, Leclere C, Renout M, Berlingo L, Cohen D, Jouannic JM. Impact of COVID-19 lockdown on maternal psychological status, the couple's relationship and mother-child interaction: a prospective study. BMC Pregnancy Childbirth. 2022 Sep 26;22(1):732. doi: 10.1186/s12884-022-05063-6. PMID 36163044